**Study Title:** A pilot cluster randomized controlled trial of a phone intervention supporting family caregivers of people living with dementia in Vietnam: Resources for Enhancing Alzheimer's Caregiver Health in Vietnam (REACH VN)

**NCT#:** NCT05481320

**Document Date:** July 14, 2022

**Document Type**: Inform Consent

## Information sheet for verbal consent – Enhanced control group

- This project is part of a research study to help us test a phone intervention to help family members who are caring for someone with memory loss or dementia.
- This study is being conducted by the National Geriatric Hospital together with researchers in the United States.
- This is a voluntary study. You are not obligated to participate. There will be no adverse consequence if you choose not to participate.
- If you agree to participate, you will receive an educational session and educational materials to help care for someone with memory loss.
- You will also meet two times over the phone to answer questionnaires about your health, well-being, and the care you provide to your relative.
- You may experience discomfort or fatigue in answering questions. Some questions may be upsetting to respond to. You can stop the interviews at any point.
- We will keep your participation in this research confidential. Your name will not appear
  in any of the records and only the research staff will have access to the data we are
  collecting.
- We will reimburse you \$8 (or 200,000 VND) at the end of each study visit.

Please contact Dr. Trong Hung Nguyen at the National Geriatric Hospital at (84) 986555666 if you have any questions.

## Information sheet for verbal consent – REACH VN Phone Intervention

- This project is part of a research study to help us test a phone intervention to help family members who are caring for someone with memory loss or dementia.
- This study is being conducted by the National Geriatric Hospital together with researchers in the United States.
- This is a voluntary study. You are not obligated to participate. There will be no adverse consequence if you choose not to participate.
- If you agree to participate, you will receive trainings from a community health worker who will meet with you during the first session at your home or another location that is convenient to you and 4-6 times over the course of 1-3 months over the phone. During our meetings, you will receive information and training to help you learn more about your relative's condition, how to provide better care, and how to improve your own health and well-being.
- You will also meet two times over the phone to answer questionnaires about your health, well-being, and the care you provide to your relative.
- You may experience discomfort or fatigue in answering questions. Some questions may be upsetting to respond to. In the intervention, some of the discussion topics may be upsetting to you. A trained interventionist (community health worker) will be able to help you should this occur. Also, you can stop at any point.
- For training purposes only, we may ask to audio record the intervention sessions. The recordings will be reviewed by a supervisor within 3 months and then destroyed. If you do not wish to have the sessions audio recorded, you may choose not to without any consequence to your study participation.
- We will keep your participation in this research confidential. Your name will not appear in any of the records and only the research staff will have access to the data we are collecting.
- We will reimburse you \$8 (or 200,000 VND) at the end of each study visit.

Please contact Dr. Trong Hung Nguyen at the National Geriatric Hospital at (84) 986555666 if you have any questions.